CLINICAL TRIAL: NCT01696227
Title: Targeted Pathogen Replacement With Novel Probiotic Treatment for Prevention of Recurrent UTIs in Children
Brief Title: Novel Probiotic Treatment for Prevention of Recurrent UTIs in Children
Acronym: Nissle 1917
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Elizabeth Lucas, Fellow MD, Nationwide Children's Hospital
Other Study IDs: IRB12-00279
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Recurrent UTIs; Catheter-Related Infections
Keywords: Nissle 1917; Probiotic; Uropathogen
MeSH Terms: conditions — Urinary Tract Infections; Catheter-Related Infections | interventions — Probiotics

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacteria recovered from samples will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nissle 1917: In vitro, Nissle 1917's ability to adversely affect the growth of uropathogens associated with urinary catheters and those with a known GI resevoir will be measured.
  Interventions: Drug: Nissle 1917

INTERVENTIONS:
Drug: Nissle 1917 — Uropathogens will be challenged to share the same in vitro environment with Nissle 1917.
  Other Names: Probiotic; Mutaflor

SUMMARY:
Background:

Urinary tract infections (UTIs) are a common and costly cause of doctor visits for children. Frequent UTIs trigger kidney damage that leads to serious diseases like high blood pressure, pregnancy complications, and kidney failure. Treating UTIs with preventative antibiotics has not shown improvement of the risk of these diseases, and contributes to the growing public health issue of antibiotic resistant bacteria. Bacteria that cause UTIs originate from the bowel. In an effort to reduce the number of UTIs, investigators want to exchange the bacteria living in our bowels for a more harmless variety.

Hypothesis and specific aims:

Investigators hypothesize a probiotic comprised of a probiotic bacteria will change the bowel bacteria, thereby reducing the numbers of infection-causing bacteria, thus reducing frequency of UTIs in healthy patients with recurrent UTIs and those patients with urinary tract problems that require use of catheters to empty their bladders.

Aim 1: Investigators plan to challenge infection-causing bacteria like Pseudomonas species, Enterococcus species, and Klebsiella species to live in the same environment with the probiotic bacteria to see how the numbers of each bacteria change.

Aim 2: Investigators will culture bacteria that live on urinary catheters and then challenge them to live in the same environment as the probiotic bacteria.

Potential Impact:

This novel treatment prevents UTIs by exchanging a patient's bowel bacteria for a harmless bacteria and reduces the use of antibiotics overall in the community.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urinary catheters placed that will be getting them removed

Exclusion Criteria:

* Patient's currently getting treated for UTI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with urinary catheters that will be getting them removed
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Ability of Nissle 1917 to adversely affect the growth in vitro of identified uropathogens | 2 years
  Uropathogens obtained from discarded clinical samples will be challenged to live in the same environment as the probiotic, Nissle 1917. Colonies of uropathogens and Nissle 1917 will be counted as a measure of the more successful organism as well as, zone of inhibition will be measured in co-cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lucas, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States